CLINICAL TRIAL: NCT05371236
Title: Development and Validation of the Spiritual Health Scale in Chinese Pediatric Cancer Patients
Brief Title: Spiritual Health Scale in Chinese Pediatric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: SPH
Record Dates: First submitted 2022-01-28; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Child
Keywords: cancer; spiritual health
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Phase I will use a descriptive qualitative approach to understand pediatric cancer patients' opinions related with spiritual issues and experience. The results of the qualitative study will be used to compare with the items of the original scale, and emerging themes will be used to generate new items. Phase Ⅱ will translates the original scale and validates the psychological properties of scale adapted for pediatric cancer patients.

SUMMARY:
Pediatric cancer patients experience spiritual concerns such as meaningless, hopeless of life, fear of death and losses at all stages of illness. The availability of a valid and reliable instrument that accurately assesses the level of spiritual health among pediatric cancer patients is crucial before any appropriate interventions to solve their spiritual concerns can be appropriately planned and evaluated.

DETAILED DESCRIPTION:
The study aimed to adapt the 12-item Functional Assessment of Chronic Illness Therapy-Spiritual Well-being Scale (FACIT-Sp-12) scale and validate it in Chinese pediatric cancer patients.

A two-phase sequential method design will be used. Phase I will use a descriptive qualitative approach to understand pediatric cancer patients' opinions related with spiritual issues and experience. At least 12 participants are expected to be interviewed. The results of the qualitative study will be used to compare with the items of the original scale, and emerging themes will be used to generate new items. Phase Ⅱ will translates and adapt the scale based on the result of Phase I. Further, the adapted version of the scale will be validated among 200 pediatric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age 8-17 years old,
* diagnosed with any type of cancer who were treated at these sites at any point after their diagnosis,
* knowing about condition and prognosis of their disease,
* their parents agree to sign the informed consent form,
* able to communicate with Chinese and read Chinese.

Exclusion Criteria:

* younger than age 8-17 years old
* cancer survivors

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The adapted spiritual well-being scale of the Functional Assessment of Chronic Illness Therapy-12 (FACIT-Sp-12) for pediatric cancer patients | past senven days
  For measuring participants' spiritual well-being
The Chinese version of the center for epidemiology studies depression scale for children (CES-DC) | past seven days
  For measuring participants' depressive symptoms
Pediatric quality of life inventory 3.0 cancer module (PedsQL 3.0 Cancer Module) | past seven days
  For measuring participants' quality of life
Socio-demographic and clinical characteristics | on that day filling out questionnaire
  For collecting the background information of the participants, including their age, gender, educational attainment, household income, number of siblings, parents' marital status and religious belief. In addition, participants' medical records will be retrieved to acquire their diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No